CLINICAL TRIAL: NCT01425905
Title: Mood and Insulin Resistance in Adolescents At-Risk for Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110239; 11-CH-0239
Record Dates: First submitted 2011-08-27; First posted 2011-08-30 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2016-01-27

CONDITIONS: Depression; Impaired Glucose Tolerance
Keywords: Female; Depression; Obesity; Insulin Resistance; Adolescents; Overweight; Type 2 Diabetes Risk; Mood
MeSH Terms: conditions — Depression; Glucose Intolerance; Obesity; Insulin Resistance; Overweight

ARMS (2):
- Depression Prevention (Experimental)
  Interventions: Other: The Blues Program
- Health Education (Active Comparator)
  Interventions: Other: Hey Durham

INTERVENTIONS:
Other: The Blues Program
  Arms: Depression Prevention
Other: Hey Durham
  Arms: Health Education

SUMMARY:
Background:

Type 2 diabetes is a chronic disease that puts individuals at risk for serious health problems like heart disease, kidney failure, vision problems, and stroke. A major way that type 2 diabetes occurs is through insulin resistance. Insulin resistance means that insulin (an important hormone in the body to keep blood sugar normal) isn t working as well as it should, which can lead to problems with high blood sugar. Insulin resistance has been linked to mood problems, stress, and depression, especially in women. To determine if group programs can help reduce the risk for type 2 diabetes, researchers want to look at teenage girls who are at risk for developing the disease.

Objectives:

To test whether a group program designed to improve mood also can help improve insulin resistance in teenage girls who are at risk for developing type 2 diabetes, or whether a group program that teaches healthy living skills is just as helpful.

Eligibility:

Teenage girls between 12 and 17 years of age who are at risk for developing type 2 diabetes.

Design:

* Participants will have two screening visits to find out if they are eligible to take part in the study. The first visit takes about 3 hours and will involve a physical exam, medical history, questionnaires and an interview about mood problems and possible depression. The second visit takes about 6 hours and will involve a full body scan to measure muscle and fat, blood draws and a glucose test to determine insulin resistance, questionnaires about general well-being and eating habits, eating meals and snacks, and an exercise test.
* Participants will join one of two group programs at the National Institutes of Health. One group focuses on learning skills to help with bad moods and stress. The other group covers topics that are important for teens to lead a healthy life. The groups will meet for 1 hour once a week for 6 weeks during after-school hours.
* At the end of the groups, participants will have three follow-up visits. The first visit will be 6 weeks later, the second will be 6 months after the start of the group program, and the third will be 1 year after the start of the group program. Each visit will take about 6 hours. These visits are similar to the second screening visit before the groups.
* Some participants will have extra tests to study stress at the second screening visit and the 6-week, 6-month, and 12-month follow-up visits. Participants will give samples of DNA, saliva to measure stress hormones, and they will take part in a brief stress test.

For more information, visit the study website at: http://mir.nichd.nih.gov or contact the research coordinators for the study at 301-594-3198.

DETAILED DESCRIPTION:
The alarming rise in prevalence of type 2 diabetes (T2D) among adolescents and young adults poses an enormous public health burden. Insulin resistance (IR) is a major physiological precursor to T2D. Depressive symptoms are associated with IR in adolescents and adults, predict adult-onset T2D, and contribute to increased risk for T2D mortality and morbidity. Depressive symptoms theoretically induce IR by promoting stress-induced behaviors (altered eating, lowered fitness) and upregulating physiological stress mechanisms (cortisol, NPY).

Psychotherapy for depression improves IR in adults, but it is unknown if ameliorating depressive symptoms prevents progression of IR in adolescents at risk for T2D. The aims of this protocol are: 1) to assess the effects of a 6-week cognitive-behavioral (CB) depression prevention group (the Blues Program) vs. a 6-week standard-of-care health education (HE) group on reducing depressive symptoms and improving IR in adolescent girls at risk for T2D; 2) to assess the stress-related behavioral and physiological factors that mediate the relationship underlying decreases in depressive symptoms and improvements in IR; and 3) to test if genotypic variation in NPY is related to severity of depressive symptoms and IR and moderates the efficacy of the CB intervention. The proposed study will permit a rigorous test of the degree to which depressive symptoms contribute to IR. The Blues Program is brief, easy-to-administer, cost-effective, and efficacious for reducing depressive symptoms among adolescent girls. If the Blues Program also improves IR, it would have the potential to have a major impact on T2D prevention in a considerable subset of youth.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 12-17 years
* Female
* BMI greater than or equal to 85th percentile for age.
* CES-D greater than or equal to 16
* Good general health
* T2D or prediabetes (impaired fasting glucose greater than or equal to 100 mg/dL or impaired glucose tolerance: 2h glucose tolerance test glucose greater than or equal to 140 mg/dL) family history in a first- or second- degree relative.
* English-speaking

EXCLUSION CRITERIA:

* Current major depressive episode
* Current psychiatric symptoms requiring treatment
* Fasting glucose >126 mg/dL
* 2-hour OGTT glucose >200 mg/dL
* Pregnancy
* Use of medication affecting IR, weight, or mood
* Current psychotherapy or weight loss treatment

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 174 (Actual)
Dates: Start 2011-08-23; Primary Completion 2015-08-10 (Actual); Study Completion 2015-08-10 (Actual)

PRIMARY OUTCOMES:
Insulin Resistance at 12 months in CB depression prevention versus HE control group.

SECONDARY OUTCOMES:
Depressive symptoms at 12 months in CB depression prevention versus HE control group.
CB, depression, prevention, group, will, show, greater, improvements, in, mediators, (eating, behavior, fitness, and stress biomarkers) than the HE control group.

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Moss SE, Klein R, Klein BE. Cause-specific mortality in a population-based study of diabetes. Am J Public Health. 1991 Sep;81(9):1158-62. doi: 10.2105/ajph.81.9.1158. PMID 1951827
- [Background] Fox CS, Coady S, Sorlie PD, D'Agostino RB Sr, Pencina MJ, Vasan RS, Meigs JB, Levy D, Savage PJ. Increasing cardiovascular disease burden due to diabetes mellitus: the Framingham Heart Study. Circulation. 2007 Mar 27;115(12):1544-50. doi: 10.1161/CIRCULATIONAHA.106.658948. Epub 2007 Mar 12. PMID 17353438
- [Background] Cheung N, Mitchell P, Wong TY. Diabetic retinopathy. Lancet. 2010 Jul 10;376(9735):124-36. doi: 10.1016/S0140-6736(09)62124-3. Epub 2010 Jun 26. PMID 20580421
- [Derived] Gulley LD, Shomaker LB, Kelly NR, Chen KY, Olsen CH, Tanofsky-Kraff M, Yanovski JA. Examining cognitive-behavioral therapy change mechanisms for decreasing depression, weight, and insulin resistance in adolescent girls at risk for type 2 diabetes. J Psychosom Res. 2022 Jun;157:110781. doi: 10.1016/j.jpsychores.2022.110781. Epub 2022 Mar 10. PMID 35367918
- [Derived] Shomaker LB, Kelly NR, Pickworth CK, Cassidy OL, Radin RM, Shank LM, Vannucci A, Thompson KA, Armaiz-Flores SA, Brady SM, Demidowich AP, Galescu OA, Courville AB, Olsen C, Chen KY, Stice E, Tanofsky-Kraff M, Yanovski JA. A Randomized Controlled Trial to Prevent Depression and Ameliorate Insulin Resistance in Adolescent Girls at Risk for Type 2 Diabetes. Ann Behav Med. 2016 Oct;50(5):762-774. doi: 10.1007/s12160-016-9801-0. PMID 27333897
- [Derived] Radin RM, Tanofsky-Kraff M, Shomaker LB, Kelly NR, Pickworth CK, Shank LM, Altschul AM, Brady SM, Demidowich AP, Yanovski SZ, Hubbard VS, Yanovski JA. Metabolic characteristics of youth with loss of control eating. Eat Behav. 2015 Dec;19:86-9. doi: 10.1016/j.eatbeh.2015.07.002. Epub 2015 Jul 18. PMID 26210388